CLINICAL TRIAL: NCT04728373
Title: An Analysis of Air-Crash Injury Patterns Presenting at a Level 1 Trauma Unit in Johannesburg, a Retrospective Cohort Study.
Status: Completed | Type: Observational
Sponsor: Sefako Makgatho Health Sciences University (Other)
Responsible Party: Principal Investigator, shumani Makhadi, Trauma Fellow, Sefako Makgatho Health Sciences University
Other Study IDs: M180463
Record Dates: First submitted 2021-01-23; First posted 2021-01-28 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Aircraft Accident
MeSH Terms: interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: surgery — the need for surgery after aircraft accidents

SUMMARY:
Aviation related deaths are often fatal, with most patients dying at the scene; however, with increased safety and improvement in medical management, patients are surviving aviation accidents. Among the aviation-related deaths reported between 1980 and 1990, polytrauma was listed as the immediate cause of death in 42% of fatalities, followed by head injuries (22%), internal organ injuries of the thorax, abdomen, pelvis (12%), burns (4%), and drowning (3%) .

Analysis and interpretation of aviation-pattern injuries may provide healthcare facilities with planning information on the spectrum of possible injuries that may be expected, and, furthermore, tools for a protocol and guidelines on the comprehensive and complete management of such patients.

The aim of the study was to describe the injury patterns, and mortality rate resulting from air crashes presenting at a level 1 trauma centre in Johannesburg, South Africa

DETAILED DESCRIPTION:
In the twenty-first century, transportation disasters and subsequent injuries are on the rise, in particular air travel, and, thus, contributing significantly to the morbidity and mortality of this millennium. However, information regarding injuries sustained by air crash survivors is lacking. As the number of commercial and non-commercial flights are increasing, health care facilities are faced with a rise in the number of patients with air crash injuries. Consequently, management guidelines must be formulated for the treatment of patients with these air crash injuries.

According to the South African Civil Aviation authority, 565 aviation accidents and incidents were reported from 2011 to 2019. The injuries and outcomes of patients involved in these accidents are unknown. There is little data to describe injury patterns and outcomes of patients in aviation accidents within our setting. Consequently, to find data on the frequency distribution of aviation injury patterns in hospitalized patients, one must use other data sources Injury patterns from several aircraft disasters have been previously described. Some authors have described injury patterns and fatalities from aviation accidents based on their patients and aircraft data. Friedman et al. described that when a plane impacts with the ground, the landing gear of an aircraft may be retracted, resulting in energy being directly transmitted from the aircraft to the passengers, through the body of the aircraft from the bottom going upwards along the axial skeleton causing vertebral column injuries that are coming with air crash patients. Therefore, it is of utmost importance that such survivors of crashes be transferred to an adequately equipped trauma center.

In 2009, Baker et al. aimed to explore the configurations of aviation-related injuries in hospitals in the United States of America (USA) whilst comparing them to the aviation deaths over the same time frame (2000 - 2005). This revealed just over 4500 aviation-related (87% non-commercial aircraft, and 7% commercial aircraft) deaths occurred in the USA - an average of 753 per year, with one death for every 1.3 hospitalizations. This represents the largest number of patients reported to date. Lower limb fractures/injuries were the most common sustained injuries, followed by head injuries, various open soft tissue wounds, upper extremity fractures/injuries, and lastly internal organ injuries. Head injuries were the cause of most fatalities. This study's case-fatality showed that 39% were due to vascular injuries, 13% due to burns, followed by 8% from head injuries.

Rautji et al. discussed the injury pattern examined in the post-mortem findings in eight occupants of a light executive jet aircraft crash. One body was severely burnt, but the other seven were intact. On serum blood toxicology, it was established that there was no carboxyhemoglobin present. Therefore, all burns were sustained post-mortem; concluding that the cause of death in all these cases was polytrauma. This evaluation found that the most commonly occurring fractures were ribs (72.3%), skull (55.1%), facial bones (49.4%), tibia (37.9%), and pelvis (36%) [9]. The common organ injuries were liver (48.1%), lung (37.6%), heart (35.6%), spleen (30.1%), and hemorrhagic cerebral and pulmonary injuries being 33.3% and 32.9%, respectively. Once again, injuries of sudden deceleration transmitted in a vertical fashion were also described, resulting in vertebral column injuries and extensive visceral damage.

A report discussed by Afshar et al. illustrated that up to 85% of injuries of survivors of a Boeing 727 flight were extremity injuries (particularly lower limb injuries), followed by vertebral column injuries at various levels, and a minority sustained internal organ injuries . Similarly, Rowles et al. (1990) concluded that most M1 Kegworth air crash injuries were orthopedic in nature, approximately 85%, and 3.8% were general surgical procedures (laparotomies, thoracotomies, vascular repair, and a tracheostomy).

Aviation related deaths are often fatal, with most patients dying at the scene; however, with increased safety and improvement in medical management, patients are surviving aviation accidents. Among the aviation-related deaths reported between 1980 and 1990, polytrauma was listed as the immediate cause of death in 42% of fatalities, followed by head injuries (22%), internal organ injuries of the thorax, abdomen, pelvis (12%), burns (4%), and drowning (3%) .

Analysis and interpretation of aviation-pattern injuries may provide healthcare facilities with planning information on the spectrum of possible injuries that may be expected, and, furthermore, tools for a protocol and guidelines on the comprehensive and complete management of such patients.

Aim of the study was to describe the injury patterns, and mortality rate resulting from air crashes presenting at a level 1 trauma centre in Johannesburg, South Africa

ELIGIBILITY:
Inclusion Criteria:

* all patients involved in aircraft accidents presenting to the hospital

Exclusion Criteria:

* patients who died on scene

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all aircraft accidents victims
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2011-01 (Actual); Primary Completion 2019-12 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
An Analysis of Air-Crash Injury Patterns Presenting at a Level 1 Trauma Unit | 8 years
  An Analysis of Air-Crash Injury Patterns Presenting at a Level 1 Trauma Unit in Johannesburg, a retrospective cohort study

SECONDARY OUTCOMES:
An Analysis of Air-Crash Injury Patterns Presenting at a Level 1 Trauma Unit in Johannesburg, a retrospective cohort study | 8 years
  28 day in-hospital mortality post aircraft accidents

CONTACTS AND LOCATIONS:
Overall Officials: Shumani Makhadi, Mmed, Principal Investigator — Sefako Makgatho Health Sciences University

IPD SHARING:
Plan to Share IPD: Undecided
protocol, study report, and statistical analysis

REFERENCES:
- [Background] Friedman A, Floman Y, Sabatto S, Safran O, Mosheiff R. Light aircraft crash--a case analysis of injuries. Isr Med Assoc J. 2002 May;4(5):337-9. PMID 12040820
- [Background] Lundin T. Transportation disasters--a review. J Trauma Stress. 1995 Jul;8(3):381-9. doi: 10.1002/jts.2490080302. No abstract available. PMID 7582604